CLINICAL TRIAL: NCT06548763
Title: Oral Topotecan in Combination With Toripalimab for Patients With Advanced/Recurrent Endometrial Cancer: a Phase II Clinical Study
Brief Title: Oral Topotecan With Toripalimab for Patients With Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Director of Gynecological Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECR-TT-2024
Record Dates: First submitted 2024-07-28; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Topotecan; Toripalimab
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Topotecan; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topotecanwith Terriptylimab (Experimental): Oral administration of topotecan and intravenous infusion of trastuzumab until disease progression or toxicity intolerance occurs.
  Interventions: Drug: Topotecan; Drug: Toripalimab

INTERVENTIONS:
Drug: Topotecan — 1.4mg/㎡, orally administered, d1-5
Drug: Toripalimab — 240mg, intravenous drip, d1, q3w

SUMMARY:
This study aims to explore the safety and efficacy of oral topotecan combined with toripalimab in treating advanced/recurrent endometrial cancer through a single-center, prospective, single-arm, phase II clinical trial. The goal is to explore the first-line treatment options for endometrial cancer patients in the era of immunotherapy, to improve the overall treatment level and prognosis of endometrial cancer.

DETAILED DESCRIPTION:
1. Overall Design This trial is a single-center, prospective, single-arm, phase II clinical trial to evaluate the safety and efficacy of oral topotecan combined with toripalimab in treating advanced/recurrent endometrial cancer.
2. Experimental observation indicators 1) Main indicators: progression-free survival (PFS), 2) Other indicators: overall survival (OS), objective response rate (ORR), adverse reactions, changes in immune-related factors and biomarkers
3. Sample size calculation This clinical trial aims to evaluate the safety and efficacy of oral topotecan combined with toripalimab in treating advanced/recurrent endometrial cancer patients. Based on literature reports, the median PFS of patients with advanced/recurrent endometrial cancer is 3.8 months. In comparison, the experimental group is expected to have a median PFS of 7 months, with an alpha value of 0.05. Follow-up for 1 year is conducted, considering a 10% dropout rate. This study plans to include 30 patients with advanced/recurrent endometrial cancer.

   Mid-term analysis: Expected ORR not less than 15%, with a minimum of 19 enrolled cases for mid-term analysis (at least 3 cases of CR or PR)
4. Methods Topotecan, 1.4mg/㎡, orally administered, d1-5+toripalimab 240mg, intravenous drip, d1, q3w, until disease progression or toxicity intolerance.
5. Data Processing Enter data and use SPSS statistical software for statistical analysis. Statistical analyst: Clinical Statistics Department of Fudan University Cancer Hospital. Mailing address: 270 Dong'an Road, Shanghai.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, female;
2. Patients with advanced/recurrent endometrial cancer diagnosed by histopathology and failed first-line treatment;
3. Can provide 10 pathological white films for subsequent research;
4. Physical fitness status score ECOG ≤ 2;
5. Expected survival period ≥ 3 months;
6. The subjects can understand the research process, voluntarily participate in this study, sign informed consent forms, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Pregnant and lactating patients, women of childbearing age who refuse to take effective contraceptive measures during the study period; Individuals with peripheral nervous system disorders caused by diseases or those with a history of significant mental and central nervous system disorders;
2. Serious or uncontrolled infections that may affect research treatment or evaluation of research results, including but not limited to active hepatitis virus infections, positive human immunodeficiency virus (HIV) antibodies, lung infections, etc;
3. Individuals who are known to be allergic, highly sensitive, or intolerant to the active ingredients or other components of the investigational drug;
4. Other malignant tumors have appeared within the past 5 years, except for cured cervical carcinoma in situ and non melanoma skin cancer;
5. Patients who are currently participating or have participated in other clinical trials within the past month;
6. The researchers determined that the patients were not suitable to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Two years
  Progression free survival

SECONDARY OUTCOMES:
OS | Two years
  Overall Survival
ORR | Two years
  Overall Remission Rate

OTHER OUTCOMES:
Tumor markers | Two years
  Substances that can reflect the occurrence and development of tumors, and monitor tumor response to treatment, including CA125, HE4, CA199, CA153, and CEA

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university shanghai cancer center, Deparment of gynecologic oncology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No